CLINICAL TRIAL: NCT01973647
Title: Efficacy and Mechanisms of a Behavioral Therapy for Insomnia Co-existing With COPD
Brief Title: A Behavioral Therapy for Insomnia Co-existing With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Mary C. Kapella, Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013-0626
Record Dates: First submitted 2013-10-22; First posted 2013-10-31 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Insomnia; COPD; Chronic Obstructive Pulmonary Disease; Fatigue
Keywords: insomnia; cognitive behavioral therapy; COPD; fatigue
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Pulmonary Disease, Chronic Obstructive; Fatigue | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cognitive Behavioral Therapy (CBT-I) (Experimental): Six weekly sessions of Cognitive Behavioral Therapy for Insomnia
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia
- CBT-I + COPD-ED (Experimental): Six weekly sessions of Cognitive Behavioral Therapy for Insomnia plus COPD Education
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia; Behavioral: COPD Education
- COPD Education (COPD-ED) (Experimental): Six weekly sessions of COPD education
  Interventions: Behavioral: COPD Education
- Attention Control (AC) (Placebo Comparator): Six weekly sessions of non-sleep, non-COPD health education
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — Six weekly sessions of cognitive behavioral therapy for insomnia
  Arms: CBT-I + COPD-ED; Cognitive Behavioral Therapy (CBT-I)
Behavioral: COPD Education — Six weekly sessions of COPD education
  Arms: CBT-I + COPD-ED; COPD Education (COPD-ED)
Behavioral: Attention Control — Six weekly sessions of non-sleep, non-COPD health education
  Arms: Attention Control (AC)

SUMMARY:
Difficulty falling asleep, staying asleep or poor quality sleep (insomnia) is common in people with chronic obstructive pulmonary disease. Insomnia is related to greater mortality, with four times the risk of mortality for sleep times < 300 minutes. Insomnia is also related to greater morbidity, with 75% greater health care costs than people without insomnia. However, insomnia medications are used with caution in COPD due to potential adverse effects. Common features of COPD such as dyspnea, chronic inflammation, anxiety and depression also affect insomnia and can interfere with therapy outcomes. While cognitive behavioral therapy for insomnia (CBT-I), a therapy that provides guidance on changing unhelpful sleep-related beliefs and behavior, is effective for people with primary insomnia and people with other chronic illnesses, the efficacy and mechanisms of action of such a therapy are yet unclear in people with both insomnia and COPD. The objective in this application is to rigorously test efficacy of two components of insomnia therapy - CBT-I and COPD education (COPD-ED) - in people with coexisting insomnia and COPD, and to identify mechanisms responsible for therapy outcomes. The central hypothesis is that both CBT-I and COPD-ED will have positive, lasting effects on objectively and subjectively measured insomnia and fatigue. The rationale for the proposed study is that once the efficacy and mechanisms of CBT-I and COPD-ED are known, new and innovative approaches for insomnia coexisting with COPD can be developed, thereby leading to longer, higher quality and more productive lives for people with COPD, and reduced societal cost due to the effects of insomnia. The investigators plan to test our central hypothesis by completing a randomized controlled comparison of CBT-I, COPD-ED and non-COPD, non-sleep health education attention control (AC) using a highly efficient 4-group design. Arm 1 comprises 6 weekly sessions of CBT-I+AC; Arm 2=6 sessions of COPD-ED+AC; Arm 3=CBT-I+COPD-ED; and Arm 4=AC. This design will allow completion of the following Specific Aims: 1. Determine the efficacy of individual treatment components, CBT-I and COPD-ED, on insomnia and fatigue. 2. Define mechanistic contributors to the outcomes after CBT-I and COPD-ED. The research proposed in this application is innovative because it represents a new and substantive departure from the usual insomnia therapy, namely by testing traditional CBT-I with education to enhance outcomes.

DETAILED DESCRIPTION:
The investigators plan to test our central hypothesis by completing a randomized controlled comparison of CBT-I, COPD-ED and non-COPD, non-sleep health education attention control (AC) using a highly efficient 4-group design. Arm 1 comprises 6 weekly sessions of CBT-I+AC; Arm 2=6 sessions of COPD-ED+AC; Arm 3=CBT-I+COPD-ED; and Arm 4=AC. This design will allow completion of the following Specific Aims: 1. Determine the efficacy of individual treatment components, CBT-I and COPD-ED, on insomnia and fatigue. 2. Define mechanistic contributors to the outcomes after CBT-I and COPD-ED.

ELIGIBILITY:
Inclusion Criteria:

* mild to very severe COPD.
* age ≥ 45 years of age with no other major healthproblems.
* clinically stable at the time of enrollment into the study.
* insomnia.

Exclusion criteria:

* evidence of restrictive lung disease or asthma.
* pulse oximetry reading of < 90% at rest or < 85% at night for > 5 min.
* evidence of a major sleep disorder other than insomnia.
* hypnotic use.
* acute respiratory infection within the previous 2 months.
* presence of a potentially debilitating disease such as cancer, congestive heart failure, kidney disease, liver failure or cirrhosis; evidence of alcohol or drug abuse, musculoskeletal or degenerative nerve disease.
* a self-reported current diagnosis of major depression or psychiatric disease or a Hospital Anxiety and Depression Scale (HADS) depression score of > 11.
* currently participating in pulmonary rehabilitation.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2014-06; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Insomnia | Up to 18 weeks
  Change in the level of insomnia will be assessed using actigraphy and the Sleep Impairment Index questionnaire.

SECONDARY OUTCOMES:
Fatigue | Up to 18 weeks
  Change in the level of fatigue will be assessed using the Chronic Respiratory Disease Questionnaire Fatigue scale and the PROMIS Fatigue scale.
Beliefs about sleep | Up to 18 weeks
  Change in beliefs about sleep will be measured using the DBAS questionnaire
Sleep habits | Up to 18 weeks
  Change in sleep habits will be measured using a Sleep Diary and Actigraphy
Self-efficacy for sleep | Up to 18 weeks
  Change in self-efficacy for sleep will be measured using the Self-efficacy for Sleep Scale
Self-efficacy for COPD management | Up to 18 weeks
  Change in self-efficacy for COPD management will be measured using the Self-efficacy for COPD scale.
Emotional arousal | Up to 18 weeks
  Change in emotional arousal will be measured using the PROMIS anxiety and depression scales
Inflammation | 6 weeks
  Change in inflammation will be measured using C-reactive protein.
Pulmonary function | 6 weeks
  Change in pulmonary function will be measured using pulmonary function tests.
Daytime functioning | Up to 18 weeks
  Change in daytime functioning will be measured using actigraphy, the Chronic Respiratory Disease Questionnaire Dyspnea Scale and the PROMIS Physical Functioning Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Mary C Kapella, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kapella MC, Herdegen JJ, Perlis ML, Shaver JL, Larson JL, Law JA, Carley DW. Cognitive behavioral therapy for insomnia comorbid with COPD is feasible with preliminary evidence of positive sleep and fatigue effects. Int J Chron Obstruct Pulmon Dis. 2011;6:625-35. doi: 10.2147/COPD.S24858. Epub 2011 Nov 24. PMID 22162648
- [Derived] Jun J, Park C, Fritschi C, Balserak B, Martyn-Nemeth P, Kuna S, Kapella M. Behavioral interventions and symptom cluster change in adults with chronic obstructive pulmonary disease and insomnia. Heart Lung. 2024 Mar-Apr;64:6-13. doi: 10.1016/j.hrtlng.2023.11.001. Epub 2023 Nov 15. PMID 37976563
- [Derived] Kapella M, Steffen A, Prasad B, Laghi F, Vispute S, Kemner G, Teixeira C, Peters T, Jun J, Law J, Carley D. Therapy for insomnia with chronic obstructive pulmonary disease: a randomized trial of components. J Clin Sleep Med. 2022 Dec 1;18(12):2763-2774. doi: 10.5664/jcsm.10210. PMID 35946416
- [Derived] Kapella MC, Herdegen JJ, Laghi F, Steffen AD, Carley DW. Efficacy and mechanisms of behavioral therapy components for insomnia coexisting with chronic obstructive pulmonary disease: study protocol for a randomized controlled trial. Trials. 2016 May 23;17(1):258. doi: 10.1186/s13063-016-1334-0. PMID 27215949